CLINICAL TRIAL: NCT00776685
Title: Cognitive Behavioral Interventions That Target Personality Risk for Substance Abuse and Mental Illness: Delivery by Educational Professionals
Brief Title: Adventure: Teacher Delivered Personality-targeted Interventions for Substance Misuse
Acronym: Adventure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Action on Addiction (Other)
Responsible Party: Dr. Patricia Conrod, Institute of Psychiatry, King's College London
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Adventure
Record Dates: First submitted 2008-10-17; First posted 2008-10-21 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-12

CONDITIONS: Alcohol Abuse; Drug Abuse; Depression; Panic Disorder; Conduct Disorder
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Depression; Panic Disorder; Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- learning to cope with your impulsivity (Experimental): Cognitive-behavioural intervention targeting impulsive personality
  Interventions: Behavioral: Personality-targeted interventions
- learning to cope with your sensation seeking (Experimental): cognitive behavioural intervention designed to help sensation seeking youth manage their need for stimulation and excitement.
  Interventions: Behavioral: Personality-targeted interventions
- learning to cope with your anxiety sensitivity (Experimental): cognitive behavioural intervention teaching anxiety sensitive youth to manager their sensitivity to threat and anxiety.
  Interventions: Behavioral: Personality-targeted interventions
- learning to manage your negative thinking (Experimental): cognitive behavioural intervention targeting pessimistic and negative thinking in hopeless youth
  Interventions: Behavioral: Personality-targeted interventions

INTERVENTIONS:
Behavioral: Personality-targeted interventions — Motivational and cognitive behavioural interventions targeting four personality profiles. 2 90 minute group sessions with personality-matched peers facilitated by a trained teacher and co-facilitator
  Other Names: Preventure, but now delivered by teachers

SUMMARY:
Several personality factors have been shown to be associated with risk for alcohol and substance misuse, and differentiate substance abusers based on clinical profile, treatment response and susceptibility to other forms of mental illness. Personality-targeted interventions have been found to have significant preventative effects on onset and growth of drinking, binge-drinking and drinking problems in adolescents attending mainstream schools (Conrod, Castellanos & Mackie, 2008). The interventions concurrently reduced personality-specific emotional and behavioural problems (Castellanos & Conrod, 2006), and prevented the onset and escalation of drug-use over a two-year period (Conrod, Castellanos-Ryan & Strang, 2010). This cluster randomised controlled trial aims to examine whether these results can be replicated when interventions are delivered by trained educational professionals. In addition, the trial will evaluate the broader impact of the programme on cigarette smoking, school attendance, academic achievement and school-wide behaviours.

DETAILED DESCRIPTION:
The Adventure study aims to examine whether educational professionals such as teachers, mentors or individuals in a pastoral role, who are trained in carrying out personality-targeted interventions will be effective in reducing problem behaviours in a group of adolescents.

20 schools in London, U.K. were recruited for the trial, and over 2000 adolescents (mean age 13.7 years) consented to participate in the survey and intervention phases of the trial. Schools were randomly assigned to control or intervention condition, and students in intervention schools who met the criteria for any of the 4 personality risk subscales of the Substance Use Risk Profile Scale (Negative Thinking, Anxiety Sensitivity, Sensation Seeking and Impulsivity) were invited to participate in a personality-targeted intervention by trained members of staff from their schools. All participants were invited to complete follow-up surveys at 6-month intervals for 2 years. The remaining 55% of low risk students in the grad were also followed to examine population-level effects of the intervention as well.

The main outcome measures of this RCT are alcohol and illicit drug outcomes. Secondary measures include mental health symptoms, risky behaviour, school attainment and attendance, and school-wide behaviours.

It is hypothesised that teacher-delivered personality-targeted interventions will have similar preventative effects on alcohol and drug use as reported by Conrod et al (2008, 2010), in addition to the personality-specific intervention effects reported by Castellanos & Conrod (2006). In addition, broader effects of the intervention on academic achievement and school-wide behaviour will be examined in this trial, both at the individual level and at the population-level.

ELIGIBILITY:
Inclusion Criteria:

* Secondary school student

Exclusion Criteria:

* None

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3190 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Binge drinking frequency | 2 years
  Frequency in the past 6 months that subject reported drinking 5 or more alcoholic beverages (4 or more for girls) on one drinking occasion.
Drinking frequency | 2 years
  Past six months frequency of drinking
drinking quantity | 2 years
  Average number of alcoholic beverages consumed on a typical drinking occasion in the past six months
Drinking problems | 2 years
  number of drinking problems reported on an abbreviated version of the Rutger's Alcohol Problem Index.
illicit drug use events | 2 years
  Time to onset of illicit drug use

SECONDARY OUTCOMES:
Emotional and behavioural problems, targeted and school-wide effects | 2 years
  Psychiatric symptoms (depression, panic anxiety, antisocial behaviours), coping skills, motives for drinking, school attendance and attainment, in-class behaviours assessed using the Strengths and Difficulties Questionnaire and the Brief Symptom Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Conrod, PhD, Study Chair — King's College London
Locations (1):
- Institute of Psychiatry, King's College London, London, United Kingdom

REFERENCES:
- [Background] Conrod PJ, Castellanos-Ryan N, Strang J. Brief, personality-targeted coping skills interventions and survival as a non-drug user over a 2-year period during adolescence. Arch Gen Psychiatry. 2010 Jan;67(1):85-93. doi: 10.1001/archgenpsychiatry.2009.173. PMID 20048226
- [Background] Conrod PJ, Castellanos N, Mackie C. Personality-targeted interventions delay the growth of adolescent drinking and binge drinking. J Child Psychol Psychiatry. 2008 Feb;49(2):181-90. doi: 10.1111/j.1469-7610.2007.01826.x. PMID 18211277
- [Background] Conrod PJ, Stewart SH, Comeau N, Maclean AM. Efficacy of cognitive-behavioral interventions targeting personality risk factors for youth alcohol misuse. J Clin Child Adolesc Psychol. 2006 Dec;35(4):550-63. doi: 10.1207/s15374424jccp3504_6. PMID 17007600
- [Result] O'Leary-Barrett M, Mackie CJ, Castellanos-Ryan N, Al-Khudhairy N, Conrod PJ. Personality-targeted interventions delay uptake of drinking and decrease risk of alcohol-related problems when delivered by teachers. J Am Acad Child Adolesc Psychiatry. 2010 Sep;49(9):954-963.e1. doi: 10.1016/j.jaac.2010.04.011. Epub 2010 Jul 31. PMID 20732631
- [Derived] O'Leary-Barrett M, Castellanos-Ryan N, Pihl RO, Conrod PJ. Mechanisms of personality-targeted intervention effects on adolescent alcohol misuse, internalizing and externalizing symptoms. J Consult Clin Psychol. 2016 May;84(5):438-52. doi: 10.1037/ccp0000082. Epub 2016 Feb 15. PMID 26881449
- [Derived] Mahu IT, Doucet C, O'Leary-Barrett M, Conrod PJ. Can cannabis use be prevented by targeting personality risk in schools? Twenty-four-month outcome of the adventure trial on cannabis use: a cluster-randomized controlled trial. Addiction. 2015 Oct;110(10):1625-33. doi: 10.1111/add.12991. Epub 2015 Jul 14. PMID 26011508
- [Derived] Conrod PJ, O'Leary-Barrett M, Newton N, Topper L, Castellanos-Ryan N, Mackie C, Girard A. Effectiveness of a selective, personality-targeted prevention program for adolescent alcohol use and misuse: a cluster randomized controlled trial. JAMA Psychiatry. 2013 Mar;70(3):334-42. doi: 10.1001/jamapsychiatry.2013.651. PMID 23344135